CLINICAL TRIAL: NCT02915250
Title: A Randomised, Double-blind, Double-dummy, Three-period Cross-over Trial to Compare Post Prandial Blood Glucose Control of BioChaperone® Combo With Humalog® Mix25 and With Simultaneous Injections of Humalog® and Lantus® in Subjects With Type 2 Diabetes
Brief Title: A Trial to Compare Post Prandial Blood Glucose Control of BioChaperone® Combo With Humalog® Mix25 and With Simultaneous Injections of Humalog® and Lantus® in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Adocia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: BC3-CT022
Record Dates: First submitted 2016-09-21; First posted 2016-09-26 (Estimated); Last update posted 2017-06-29 (Actual); Status verified 2017-06

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Lispro; Insulin Glargine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- BioChaperone® Combo (Experimental): Individualised single subcutaneous of BioChaperone® Combo + injection of placebo (0.9% NaCl) to ensure the double dummy
  Interventions: Drug: BioChaperone® Combo; Drug: Placebo
- Humalog® Mix25 (Active Comparator): Individualised single subcutaneous of Humalog® Mix25 + injection of placebo (0.9% NaCl) to ensure the double dummy
  Interventions: Drug: Humalog® Mix25; Drug: Placebo
- Humalog® and Lantus® (Active Comparator): Individualised simultaneous subcutaneous injections
  Interventions: Drug: Humalog®; Drug: Lantus®

INTERVENTIONS:
Drug: BioChaperone® Combo — Injection of BioChaperone® Combo
  Arms: BioChaperone® Combo
Drug: Humalog® Mix25 — Injection of Humalog® Mix25
  Arms: Humalog® Mix25
Drug: Humalog® — Injection of Humalog®
  Arms: Humalog® and Lantus®
Drug: Lantus® — Injection of Lantus®
  Arms: Humalog® and Lantus®
Drug: Placebo — Injection of 0.9% NaCl
  Arms: BioChaperone® Combo; Humalog® Mix25

SUMMARY:
This is a two-centre, randomised, double-blind, double-dummy, 3-treatment, 3-period cross-over study using a standardised solid meal test in subjects with type 2 diabetes to investigate postprandial glucose control of BioChaperone® Combo compared with Humalog® Mix25 and with simultaneous subcutaneous injections of Humalog® and Lantus® during three separate dosing visits.

DETAILED DESCRIPTION:
This is a two-centre, randomised, double-blind, double-dummy, 3-treatment, 3-period cross-over study using a standardised solid meal test in subjects with type 2 diabetes to investigate postprandial glucose control of BioChaperone® Combo compared with Humalog® Mix25 and with simultaneous subcutaneous injections of Humalog® and Lantus® during three separate dosing visits.

Furthermore, this study aims to compare the pharmacokinetic (PK) profiles of the three different study treatments.

During each dosing visit, subjects will be given 3 doses of IMP on three consecutive days (Day 1, Day 2 and Day 3). Dosing on Day 2 and Day 3 will be followed by a standardised solid meal test.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject aged 18-70 years (both inclusive)
* Type 2 diabetes mellitus (as diagnosed clinically) for ≥ 12 months
* HbA1c level between 7.5% and 9.5% (both inclusive)
* Body mass index between 20.0 and 40.0 kg/m2 (both inclusive)
* Treated with once daily injections with insulin glargine U-100 for ≥ 3 months prior to screening

Exclusion Criteria:

* Type 1 diabetes mellitus
* Known or suspected allergy to the IMPs or related products
* Previous participation in this trial. Participation is defined as randomised.
* Receipt of any medicinal product in clinical development within 60 days prior to this trial.
* Clinically significant abnormal haematology, biochemistry, urinalysis or coagulation screening tests, as judged by the Investigator considering the underlying disease
* Supine blood pressure at screening outside the range of 90-160 mmHg for systolic or 50-95 mmHg for diastolic and/or resting supine heart rate outside the range 50-90 beats per minute. This exclusion criterion also pertains to subjects being on antihypertensives.
* Current treatment with premixed or intermediate insulin products, or with long acting insulins other than insulin glargine U-100. The use of short or rapid acting prandial insulin products will be allowed provided their use has been stable for ≥ 3 months prior to screening.
* Use of GLP-1 receptor agonists or oral antidiabetic drugs (OADs) other than stable intake of metformin alone or metformin in combination with a DPP-4 inhibitor within 4 weeks prior to screening
* Women of child bearing potential not willing to use contraceptive methods.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Delta AUC BG 0-2h (area under the blood glucose concentration-time curve) | From 0 to 2 hours
  Mean of incremental areas under the blood glucose concentration-time curve from 0-2 hours after a standardised meal on Day 2 and Day 3

SECONDARY OUTCOMES:
Partial delta AUCs BG and total AUCs BG | From 0 to 6 hours
  Partial incremental AUCs BG and total AUCs BG in the 0-6 time range
Mean and mean change from baseline of blood glucose at different time points | From 0 to 6 hours
Delta BGmax and delta BGmin | From 0 to 6 hours
  Maximum and minimum blood glucose excursions after a standardised meal
BGmax and BGmin | From 0 to 6 hours
  Maximum and minimum blood glucose concentrations after a standardised meal
AUC Insulin | From 0 to 24 hours
  Partial areas under the insulins plasma concentration time curve
Cmax Insulin | From 0 to 6 hours
  Maximum observed plasma insulins concentration
tmax Insulin | From 0 to 6 hours
  Time to maximum observed plasma insulins concentration
Adverse Events | Up to 12 weeks (maximum duration of subject's participation)
Local tolerability | Up to 12 weeks (maximum duration of subject's participation)
Hypoglycaemic events | Up to 12 weeks (maximum duration of subject's participation)

CONTACTS AND LOCATIONS:
Overall Officials: Leona Plum-Mörschel, MD, Principal Investigator — Profil Mainz GmbH & Co KG
Locations (2):
- Germany (2):
  - Profil Mainz GmbH & Co.KG, Mainz
  - Profil GmbH, Neuss

IPD SHARING:
Plan to Share IPD: No